CLINICAL TRIAL: NCT05273008
Title: Risk Factors for the Development of Groin Pain in Roller Hockey Athletes
Brief Title: Adductor Strength in Roller Hockey Athletes
Status: Completed | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Hugo Olmedillas Fernandez, Associate professor, University of Oviedo
Other Study IDs: UO2021-03
Record Dates: First submitted 2022-02-28; First posted 2022-03-10 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Groin Pain
Keywords: Roller hockey; Groin Pain; Risk factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active hockey players: Observational study on 180 Hockey players

SUMMARY:
Roller hockey athletes will be recruited along the season and will be examined for adductor strength and other potential groin pain risk factors.

DETAILED DESCRIPTION:
Roller hockey athletes will be recruited and assess through the season. The assessment consist of an adductor, abductor strength measurement, Hip and Groin Outcome Score (HAGOS) completion and will be screened for other risk factors which are believed to cause groin pain (Age, previous injury)

ELIGIBILITY:
Inclusion Criteria:

* Participate in the roller hockey bronze division from spain

Exclusion Criteria:

* Deny participation

Ages: 16 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Athletes playing in the spanish roller hockey´s third division
Sampling Method: Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Adductor Strength | November 2021-March 2022
  Adductor strength will be measured with a dynamometer
Abductor strength | November 2021-March 2022
  Abductor strength will be measured with a dynamometer
Adductor to abductor ratio | November 2021-March 2022
  Ratio between adductor and abductor strength will be calculated

SECONDARY OUTCOMES:
Hip and Groin Outcome Score | November 2021-March 2022
  a questionnaire will be given to every participant to obtain information on groin pain symptoms in the last week
5 seconds squeeze test | November 2021-March 2022
  While measuring adductor and abductor strength, pain will be assess during the test

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Olmedillas, PhD, Principal Investigator — Universidad de Oviedo
Locations (1):
- Universidad de Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Characterising groin pain in rink hockey: Function and five-second squeeze in Spanish players — https://doi.org/10.1016/j.ptsp.2022.10.004